CLINICAL TRIAL: NCT05766592
Title: Affirmative Family and Individual Psychotherapy for Sexual and Gender Minority Adults and Their Nonaccepting Parents
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Ben-Gurion University of the Negev (Other); Israel Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000034163
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Mental Health Issue; Parent-Child Relations
Keywords: LGBTQ; Cognitive Behavioral Therapy; Attachment-Based Family Therapy

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be immediately assigned to either condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LGBTQ-affirmative CBT (Experimental): Individuals assigned to LGBTQ-affirmative cognitive behavioral therapy will receive 16 weekly individually-delivered sessions, directly after baseline assessment, delivered via telehealth. Based on the Unified Protocol, sessions will address minority stress mechanisms underlying sexual and gender minority mental health disparities.
  Interventions: Behavioral: LGBTQ-affirmative CBT
- ABFT-SGM (Experimental): Individuals assigned to attachment-based family therapy for sexual and gender minorities will receive a 16-session sequence of family-based therapy delivered via telehealth. This sequence will include sessions with sexual and/or gender minority adult children alone, adult children and parent(s), and parent(s) alone. Sessions will address the quality parent-child relationship in relation to child sexual orientation and gender identity to target mental health disparities.
  Interventions: Behavioral: ABFT-SGM

INTERVENTIONS:
Behavioral: LGBTQ-affirmative CBT — 16-session LGBTQ-affirmative psychotherapy using cognitive behavioral techniques
  Arms: LGBTQ-affirmative CBT
Behavioral: ABFT-SGM — 16-session attachment-based family therapy for sexual and gender minority young adults and their nonaccepting parents
  Arms: ABFT-SGM

SUMMARY:
The purpose of this study is to assess the efficacy of an LGBTQ-affirmative individual cognitive behavioral psychotherapy (CBT) and LGBTQ-affirmative family therapy (attachment-based family therapy for sexual and gender minority young adults; ABFT-SGM) delivered via telehealth to a sample of sexual and gender minority adults with nonaccepting parent(s) in New York, Pennsylvania, Connecticut, and Israel. The investigators will assess whether both treatments are associated with significant decreases in depressive and anxiety symptoms. The investigators will also assess whether and how each treatment achieves reductions in mental health symptoms through specific mechanisms (e.g., rejection sensitivity, internalized stigma, emotion dysregulation, parental rejection and acceptance).

DETAILED DESCRIPTION:
The purpose of this study is to assess the efficacy and purported change mechanisms in an LGBTQ-affirmative individual cognitive behavioral psychotherapy (CBT) and LGBTQ-affirmative family therapy (attachment-based family therapy for sexual and gender minority young adults; ABFT-SGM) delivered via telehealth to a sample of sexual and gender minority adults in New York, Pennsylvania, Connecticut, and Israel. In this 2-arm randomized clinical trial (RCT), participants will receive 16 weekly sessions of either LGBTQ-affirmative CBT or ABFT-SGM. Investigators will assess whether both treatments are associated with significant decreases in depressive and anxiety symptoms. Investigators will also assess whether psychosocial mechanisms (e.g., rejection sensitivity, internalized stigma, emotion dysregulation, parental rejection and acceptance) mediate reductions in psychological symptoms, and whether such mediators differ between the two treatments. Finally, investigators will assess whether participants who begin treatment with higher levels of parental rejection benefit more from ABFT-SGM than from LGBTQ-affirmative CBT, and whether participants with higher initial levels of maladaptive stress responses benefit more from LGBTQ-affirmative CBT.

ELIGIBILITY:
Inclusion Criteria:

* be 20 and older
* be fluent in English
* self-identify as lesbian, bisexual, queer, pansexual, or other non-heterosexual identity
* currently experience elevated depressive or anxiety symptoms (screened initially using a cutoff of ≥ 2.5 on the Brief Symptom Inventory-4 and further confirmed by the BDI and BAI).
* report at least moderate levels of parental rejection or low levels of parental acceptance, as measured using the PARSOS.
* have at least one rejecting/nonaccepting parent that agrees to participate in the therapy.
* live in New York State, Pennsylvania, Connecticut, or Israel.

Exclusion Criteria:

* report current mental health treatment ≥1 day/month (except for medication management ≤1 day/week)
* report beginning a new medication within the past 30 days
* exhibit active psychosis or active mania, as assessed by the SCID-Psych Screen.
* exhibit active suicidality or active homicidality, as assessed by the SIDAS
* be currently legally mandated to attend treatment
* demonstrate gross cognitive impairment, as assessed with the Telephone Interview for Cognitive Status
* do not have a parent willing to participate

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in depression symptoms | Baseline, Immediate Post-intervention, 5-month Post-intervention
  Depressive symptoms will be measured using the 21-item Beck Depression Inventory-II (BDI). Items are rated on a scale from 0-3 where higher scores indicate greater depression symptoms, with a maximum score of 63.
Change in anxiety symptoms | Baseline, Immediate Post-intervention, 5-month Post-intervention
  Anxiety symptoms will be measured using the 21-item Beck Anxiety Inventory (BAI). Items are rated on a scale from 0-3 where higher scores indicate greater anxiety symptoms, with a maximum score of 63.

SECONDARY OUTCOMES:
Change in suicidal ideation | Baseline, Immediate Post-intervention, 5-month Post-intervention
  Suicidal ideation will be measured using a single item from the Patient Health Questionnaire-9. This item is rated from 0-3, where a higher score indicates higher suicidal ideation.
Change in sexual orientation and gender modality concealment motivation, as relevant | Baseline, Immediate Post-intervention, 5-month Post-intervention
  Motivation to conceal sexual orientation and gender modality will be assessed using the Concealment Motivation subscale of the Lesbian, Gay, and Bisexual Identity Scale (LGBIS). The three subscale items, rated on a 6-point scale, will be averaged for a maximum total score of 6. Higher scores indicate higher concealment motivation.
Change in sexual orientation and gender modality acceptance concerns, as relevant | Baseline, Immediate Post-intervention, 5-month Post-intervention
  Acceptance concerns of sexual minority identity and gender identity will be assessed using the Acceptance Concerns subscale of the Lesbian, Gay, and Bisexual Identity Scale (LGBIS). The three subscale items, rated on a 6-point scale, will be averaged for a maximum total score of 6. Higher scores indicate higher acceptance concerns.
Change in explicit internalized stigma | Baseline, Immediate Post-intervention, 5-month Post-intervention
  Change in explicit internalized stigma will be assessed using the Internalized Homonegativity subscale of the Lesbian, Gay, and Bisexual Identity Scale (LGBIS). The three subscale items, rated on a 6-point scale, will be averaged for a maximum total score of 6. Higher scores indicate higher acceptance concerns.
Change in emotion dysregulation | Baseline, Immediate Post-intervention, 5-month Post-intervention
  Emotion dysregulation will be assessed using the 18-item Difficulties in Emotion Regulation Scale-Short Form (DERS-SF). Items are rated on a 5-point scale from 1-5; items 1, 4, and 6 are reverse coded. Items are averaged for a total maximum score of 5, where higher scores indicate higher emotion dysregulation.
Change in implicit sexual orientation bias | Baseline, Immediate Post-intervention
  Implicit bias related to sexual orientation will be measured using the sexual orientation Implicit Association Test. Scores range from -2 to 2, where higher scores indicate higher implicit preference towards heterosexuality.
Change in parental acceptance of sexual orientation or gender modality, as relevant | Baseline, Immediate Post-intervention, 5-month Post-intervention
  Parental acceptance will be measured by the Parental Acceptance subscale of the Parental Acceptance and Rejection of Sexual Orientation and Gender Identity Scale (PARSOS). 15 items are rated on a 5-point scale from 1-5. Items are averaged for a maximum total score of 5, indicating higher parental acceptance.
Change in parental rejection of sexual orientation or gender modality, as relevant | Baseline, Immediate Post-intervention, 5-month Post-intervention
  Parental rejection will be measured by the Parental Rejection subscale of the Parental Acceptance and Rejection of Sexual Orientation and Gender Identity Scale (PARSOS). 13 items are rated on a 5-point scale from 1-5. Items are averaged for a maximum total score of 5, indicating higher parental rejection.
Change in quality of attachment relationship | Baseline, Immediate Post-intervention, 5-month Post-intervention
  Quality of attachment relationship will be assessed using the Experience in Close Relationships-Relationship Structures Questionnaire (ECR-RS). 9 items are rated on a scale from 1-7 and averaged for a total maximum score of 7, indicating a higher quality of attachment relationship.

CONTACTS AND LOCATIONS:
Overall Officials: John E Pachankis, PhD, Principal Investigator — Yale University; Gary M Diamond, PhD, Principal Investigator — Ben-Gurion University of the Negev
Locations (2):
- Yale LGBTQ Mental Health Initiative with the Yale School of Public Health Office, New York, New York, United States
- Ben-Gurion University Psychotherapy Research Lab, Beersheba, Israel

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be made available to qualified researchers upon request to the PIs following study conclusion.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available 12 months after study completion for three years.
Access Criteria: Data access requests from qualified academic investigators for non-commercial research interests will be reviewed by study investigators. Requestors will be required to sign a data access agreement.

REFERENCES:
- [Background] Wang YP, Gorenstein C. Psychometric properties of the Beck Depression Inventory-II: a comprehensive review. Braz J Psychiatry. 2013 Oct-Dec;35(4):416-31. doi: 10.1590/1516-4446-2012-1048. Epub 2013 Dec 23. PMID 24402217
- [Background] Beck AT, Epstein N, Brown G, Steer RA. An inventory for measuring clinical anxiety: psychometric properties. J Consult Clin Psychol. 1988 Dec;56(6):893-7. doi: 10.1037//0022-006x.56.6.893. No abstract available. PMID 3204199
- [Background] Mohr JJ, Kendra MS. Revision and extension of a multidimensional measure of sexual minority identity: the Lesbian, Gay, and Bisexual Identity Scale. J Couns Psychol. 2011 Apr;58(2):234-245. doi: 10.1037/a0022858. PMID 21319899
- [Background] Gouveia P, Ramos C, Brito J, Almeida TC, Cardoso J. The Difficulties in Emotion Regulation Scale - Short Form (DERS-SF): psychometric properties and invariance between genders. Psicol Reflex Crit. 2022 May 6;35(1):11. doi: 10.1186/s41155-022-00214-2. PMID 35522349
- [Background] Kibrik EL, Cohen N, Stolowicz-Melman D, Levy A, Boruchovitz-Zamir R, Diamond GM. Measuring Adult Children's Perceptions of Their Parents' Acceptance and Rejection of Their Sexual Orientation: Initial Development of the Parental Acceptance and Rejection of Sexual Orientation Scale (PARSOS). J Homosex. 2019;66(11):1513-1534. doi: 10.1080/00918369.2018.1503460. Epub 2018 Aug 24. PMID 30142289
- [Background] Kasch KL, Klein DN, Lara ME. A construct validation study of the Response Styles Questionnaire Rumination Scale in participants with a recent-onset major depressive episode. Psychol Assess. 2001 Sep;13(3):375-83. doi: 10.1037//1040-3590.13.3.375. PMID 11556274
- [Background] Steffens MC, Buchner A. Implicit Association Test: separating transsituationally stable and variable components of attitudes toward gay men. Exp Psychol. 2003;50(1):33-48. doi: 10.1027//1618-3169.50.1.33. PMID 12629959
- [Background] Fraley RC, Heffernan ME, Vicary AM, Brumbaugh CC. The Experiences in Close Relationships-Relationship Structures questionnaire: a method for assessing attachment orientations across relationships. Psychol Assess. 2011 Sep;23(3):615-25. doi: 10.1037/a0022898. PMID 21443364
- [Background] Tolin DF, Gilliam C, Wootton BM, Bowe W, Bragdon LB, Davis E, Hannan SE, Steinman SA, Worden B, Hallion LS. Psychometric Properties of a Structured Diagnostic Interview for DSM-5 Anxiety, Mood, and Obsessive-Compulsive and Related Disorders. Assessment. 2018 Jan;25(1):3-13. doi: 10.1177/1073191116638410. Epub 2016 Mar 17. PMID 26988404
- [Background] Lang AJ, Norman SB, Means-Christensen A, Stein MB. Abbreviated brief symptom inventory for use as an anxiety and depression screening instrument in primary care. Depress Anxiety. 2009;26(6):537-43. doi: 10.1002/da.20471. PMID 19016462
- [Background] Cook SE, Marsiske M, McCoy KJ. The use of the Modified Telephone Interview for Cognitive Status (TICS-M) in the detection of amnestic mild cognitive impairment. J Geriatr Psychiatry Neurol. 2009 Jun;22(2):103-9. doi: 10.1177/0891988708328214. PMID 19417219
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941